CLINICAL TRIAL: NCT01906918
Title: Evaluation of Remote Preconditioning on Heart Resistance to Ischemia and Reperfusion Injury
Brief Title: Application of Remote Ischemic Preconditioning in Patients Undergoing Open Heart Surgeries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Orlando Petrucci, Phd, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RIPC
Record Dates: First submitted 2013-07-21; First posted 2013-07-24 (Estimated); Last update posted 2013-11-28 (Estimated); Status verified 2013-11

CONDITIONS: Coronary Artery Disease; Valvular Heart Disease
Keywords: ischemia; reperfusion; myocardial ischemia; myocardial reperfusion
MeSH Terms: conditions — Coronary Artery Disease; Heart Valve Diseases; Ischemia; Myocardial Ischemia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- IRPC, Remote preconditioning (Experimental): This group will be submitted to ischemic preconditioning
  Interventions: Procedure: IRPC, Remote preconditioning
- Control (Placebo Comparator): This patients will be submitted to the standard surgery protocol in the institution. The patients will not be submitted to 5 minutes of upper limb compression by cuff followed by 5 minutes of reperfusion.

INTERVENTIONS:
Procedure: IRPC, Remote preconditioning — The patients will be submitted to 5 minutes of upper limb compression by cuff followed by 5 minutes of reperfusion. This cycle will be repeated 4 times.
  Arms: IRPC, Remote preconditioning

SUMMARY:
Strategies for myocardial protection during open heart surgeries are desired. Several experimental studies have shown beneficial effects of remote ischemic preconditioning (RIPC). The underlying mechanisms are not totally understood. This study intends to evaluate molecular mechanisms involved with RIPC on myocardium of patients underwent open heart surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Scheduled for coronary artery bypass grafting with or without valve replacement associated
* Use of blood cardioplegia
* EuroSCORE II greater than or equal to 1.0%

Exclusion Criteria:

* History of cardiogenic shock
* Complications in the admission
* Pregnant patients
* Severe peripheral arterial disease affecting the upper limbs
* Liver failure (bilirubin ˃ 20 mmol / L, INR 2.0 ˃)
* Significant pulmonary disease (˂ FEV1 40%)
* Renal failure with glomerular filtration rate ˂ ml/min/1,73 m²
* Concomitant treatment with glibenclamide or nicorandil (medications that interfere with cardioprotection induced by IPCR)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-08; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Molecular pathway activation | 2 days
Inflammatory response | 10 days

SECONDARY OUTCOMES:
All cause of mortality | 30 days
All cause of mortality | 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Orlando Petrucci, MD, PhD, Study Chair — University of Campinas; Fany Lima, RN, Principal Investigator — University of Campinas
Locations (1):
- Hospital das Clínicas da Unicamp, Campinas, São Paulo, Brazil